CLINICAL TRIAL: NCT03113877
Title: Evaluation of Autonomic Function in Individuals With Cornelia de Lange Syndrome (CdLS), a Pilot Study.
Brief Title: Evaluation of Autonomic Function in Individuals With Cornelia de Lange Syndrome (CdLS)
Status: Terminated | Type: Observational
Why Stopped: Difficulty in recruitment, Funding has run out.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amie E. Jones, M.D., PI, Mayo Clinic
Other Study IDs: 15-003782
Record Dates: First submitted 2016-11-16; First posted 2017-04-14 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Cornelia de Lange Syndrome
MeSH Terms: conditions — De Lange Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clinical Testing for Autonomic Dysfunction: COMPASS-31 Survey completion. Autonomic Reflex Screen. Thermoregulatory Swear Test.
  Interventions: Other: Autonomic Dysfunction Testing

INTERVENTIONS:
Other: Autonomic Dysfunction Testing — The participants with CdLS will complete the COMPASS-31 survey and will complete standard clinical testing for autonomic dysfunction including an autonomic reflex screen (tilt table and quantitative sudomotor axon reflex testing) and thermoregulatory sweat test (TST).

SUMMARY:
Based on survey data, individuals with Cornelia de Lange Syndrome (CdLS) often experience symptoms of autonomic dysfunction however there are no reported studies in which these patients have had objective testing of the autonomic nervous system. This is a pilot study in which patients with CdLS will undergo the standard clinical testing for autonomic dysfunction with a autonomic reflex screen and thermoregulatory sweat test.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (aged 8-17 years of age) with Cornelia de Lange syndrome.
* Consent obtained from responsible guardian.

Exclusion Criteria:

* Patients less than age 8 or 18 and older
* Female patients known to be pregnant
* Individuals not thought to be able to tolerate the testing.
* Concomitant therapy with anticholinergic, alpha-adrenergic antagonists, beta-adrenergic antagonists or other medications which could interfere with autonomic testing. Patients may participate if the potentially interfering medication is held for five half-lives prior to the study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with CDLS reached through national distribution list through the CdLS Foundation with an invitation to volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-08; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who tolerated 70 degree head up tilt table test | 1 year
  Patients tolerating at least 5 minutes of tilt table
Number of patients who show evidence of dysautonomia | 1 year
  Dysautonomia measured by excessive heart rate (>40 bpm) on a tilt table test or reduced sweating on a thermoregulatory sweat test.
Number of patients who tolerated thermoregulatory sweat test | 1 year
  Patients tolerating at least 15 minutes of thermoregulatory sweat test

CONTACTS AND LOCATIONS:
Overall Officials: Amie E Jones, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No